CLINICAL TRIAL: NCT00903084
Title: A Phase 1 Pharmacokinetic Study of Varying Dosing Patterns on Tenofovir Concentrations in Hair
Brief Title: Examining Hair to Determine Tenofovir Exposure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Albert Liu, Director, HIV Prevention Intervention Studies SFDPH/Bridge HIV, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R21MH085598 (NIH); R21MH085598 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: HIV
Keywords: Pharmacokinetics in Hair; Tenofovir; Pharmacokinetics; Concentrations; Hair
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): Participants will receive 7 doses per week, then 4 doses per week, then 2 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- 2 (Active Comparator): Participants will receive 7 doses per week, then 2 doses per week, then 4 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- 3 (Active Comparator): Participants will receive 4 doses per week, then 7 doses per week, then 2 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- 4 (Active Comparator): Participants will receive 4 doses per week, then 2 doses per week, then 7 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- 5 (Active Comparator): Participants will receive 2 doses per week, then 7 doses per week, then 4 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- 6 (Active Comparator): Participants will receive 2 doses per week, then 4 doses per week, then 7 doses per week (each for 6 weeks) of tenofovir, with a break in between dosing periods.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — 300-mg tablet
  Other Names: Viread; Tenofovir

SUMMARY:
This study will determine whether a hair test can reveal how much of the anti-HIV medication tenofovir a person without HIV has been exposed to.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) is a new strategy for the prevention of HIV infection. It involves providing antiretroviral medications-those that treat HIV infections-to people before they are exposed to HIV. In clinical trials of PrEP, several of which are currently under way, accurate measurements are needed of how much exposure participants have to the PrEP medications. Current methods, such as self-reports of medication adherence or pill counting, can lead to inaccurate readings of PrEP exposure because participants may forget to take pills and individual differences may affect levels of exposure. Measuring PrEP exposure levels in hair yields an objective marker of exposure that is not subject to self-report errors and that takes into account individual differences. This study will test the use of a hair sample for assessing the level of exposure to tenofovir disoproxil fumarate (TDF), an antiretroviral medication, in people not infected with HIV.

Participation in this study will last 9 months. Participants will undergo baseline testing and then will be randomly assigned to begin one of three conditions, based on dosing schedule: receiving TDF 2, 4, or 7 days per week. All participants will complete each of these dosing schedules, but the order in which they are completed will be randomly assigned. Each dosing schedule will last 6 weeks, with a break of several weeks between them. During each dosing schedule, study staff will confirm that participants are taking each scheduled dose by watching them take the pills on weekdays and calling them on weekends. Follow-up visits will occur at Days 1, 21, and 42 of each dosing schedule. During the baseline and follow-up visits, the following will be completed: an HIV rapid test; counseling about HIV prevention; a brief physical exam; a talk with a staff member about health, symptoms, and other medications; a blood draw, which will be used for several tests; collection of a urine sample and pregnancy test; and optional donation of a sample of pubic hair. On the last day of each dosing schedule, a small sample of hair will be cut from each participant's scalp. An additional follow-up visit will occur after participants complete 4 weeks of the 7-day dosing schedule. This visit will last 24 hours and will involve collection of additional blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak English
* HIV-1 uninfected, based on HIV rapid testing performed during screening and enrollment
* Calculated creatinine clearance greater than or equal to 60 mL/min by the Cockcroft-Gault creatinine clearance formula
* Serum creatinine less than or equal to the site laboratory upper limit of normal
* Urine dipstick with negative or trace result for both glucose and protein
* Negative urine beta human chorionic gonadotropin (beta-HCG) test for women
* Adequate hepatic function, defined as total bilirubin and hepatic transaminases (ALT and AST) less than or equal to twice the upper limit of normal
* Adequate hematologic function, defined as an absolute neutrophil count greater than or equal to 1,500/mm3, platelet count greater than or equal to 100,000/mm3, and hemoglobin greater than or equal to 10 g/dL
* Ability to participate in modified directly observed dosing of study drug
* Ability to provide a personal cell phone number to be contacted on for unobserved modified directly observed therapy (mDOT) visits
* Minimum length of 3 cm scalp hair in occipital region
* Willing to provide hair and plasma samples as specified by the protocol
* Dark hair (brown or black), as assessed by the study clinician
* Volunteers born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last protocol visit for sexual activity that could lead to pregnancy and agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last scheduled protocol visit.

Exclusion Criteria:

* Active and serious medical problems, including heart or lung disease, diabetes requiring hypoglycemia medications, previously diagnosed malignancies expected to require further treatment, and serious infections
* Hepatitis B surface antigen positivity
* History of chronic kidney disease
* Known osteoporosis, osteomalacia, or osteopenia
* History of pathological bone fractures not related to trauma
* Receiving ongoing therapy with any of the following: antiretroviral therapy, interferon or interleukin therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, systemic chemotherapeutic agents, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), or other investigational agents
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting that may confer an inability to receive an orally administered medication
* Use of hair dyes or hair permanent products in the last 3 months (streaking is acceptable)
* Current participation in any other research study involving drugs, investigational agents, or medical devices
* Breastfeeding at screening or enrollment, per participant report
* Active alcohol or drug use considered sufficient by clinician to hinder compliance with study procedures
* Elevated risk of HIV infection, as defined in the study protocol
* At enrollment, has any social or medical condition that, in the investigator's opinion, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Tenofovir hair concentration under each dosing condition | Measured 6 weeks after starting each dosing condition

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Study Chair — San Francisco Department of Public Health
Locations (2):
- United States (2):
  - San Francisco Department of Public Health, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Gandhi M, Ameli N, Bacchetti P, Gange SJ, Anastos K, Levine A, Hyman CL, Cohen M, Young M, Huang Y, Greenblatt RM; Women's Interagency HIV Study (WIHS). Protease inhibitor levels in hair strongly predict virologic response to treatment. AIDS. 2009 Feb 20;23(4):471-8. doi: 10.1097/QAD.0b013e328325a4a9. PMID 19165084
- [Background] Huang Y, Gandhi M, Greenblatt RM, Gee W, Lin ET, Messenkoff N. Sensitive analysis of anti-HIV drugs, efavirenz, lopinavir and ritonavir, in human hair by liquid chromatography coupled with tandem mass spectrometry. Rapid Commun Mass Spectrom. 2008 Nov;22(21):3401-9. doi: 10.1002/rcm.3750. PMID 18837069
- [Background] Gandhi M, Greenblatt RM. Hair it is: the long and short of monitoring antiretroviral treatment. Ann Intern Med. 2002 Oct 15;137(8):696-7. doi: 10.7326/0003-4819-137-8-200210150-00016. No abstract available. PMID 12379072
- [Result] Liu AY, Yang Q, Huang Y, Bacchetti P, Anderson PL, Jin C, Goggin K, Stojanovski K, Grant R, Buchbinder SP, Greenblatt RM, Gandhi M. Strong relationship between oral dose and tenofovir hair levels in a randomized trial: hair as a potential adherence measure for pre-exposure prophylaxis (PrEP). PLoS One. 2014 Jan 8;9(1):e83736. doi: 10.1371/journal.pone.0083736. eCollection 2014. PMID 24421901
- [Result] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- See also: Click here for the San Francisco Department of Public Health HIV Research Section — http://helpfighthiv.org